CLINICAL TRIAL: NCT03492580
Title: Comparison of Canagliflozin vs. Alternative Antihyperglycemic Treatments on Risk of Heart Failure Hospitalization and Amputation for Patients With Type 2 Diabetes Mellitus and the Subpopulation With Established Cardiovascular Disease
Brief Title: A Study for Comparison of Canagliflozin Versus Alternative Antihyperglycemic Treatments on Risk of Heart Failure Hospitalization and Amputation for Participants With Type 2 Diabetes Mellitus and the Subpopulation With Established Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108464; RRA-20250 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Canagliflozin; empagliflozin; dapagliflozin; Glucagon-Like Peptide 1; Thiazolidinediones; Sulfonylurea Compounds; Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Cohort 1: Canagliflozin: A target cohort which includes new users of canagliflozin for clinical characterization, and population-level effect estimation. It will use 4 databases: 1. Truven Health MarketScan Commercial Claims and Encounters Database (CCAE) 2. Truven Health MarketScan Medicare Supplemental and Coordination of Benefits Database (MDCR) 3. Truven Health MarketScan Multi-state Medicaid Database (MDCD) 4. OptumInsight's de-identified Clinformatics Datamart, Extended-Date of Death (Optum).
  Interventions: Drug: Canagliflozin
- Cohort 2: Canagliflozin with Cardiovascular Disease (CVD): A target cohort which includes new users of canagliflozin with established CVD for clinical characterization and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Canagliflozin
- Cohort 3: Empagliflozin: A comparator cohort which includes new users of empagliflozin for clinical characterization, and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Empagliflozin
- Cohort 4: Empagliflozin with CVD: A comparator cohort which includes new users of empagliflozin with established CVD for clinical characterization and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Empagliflozin
- Cohort 5: Dapagliflozin: A comparator cohort which includes new users of dapagliflozin for clinical characterization, and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Dapagliflozin
- Cohort 6: Dapagliflozin with CVD: A comparator cohort which includes new users of dapagliflozin with established CVD for clinical characterization and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Dapagliflozin
- Cohort 7: Empagliflozin or Dapagliflozin: A target cohort which includes new users of empagliflozin or dapagliflozin for clinical characterization, and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Empagliflozin; Drug: Dapagliflozin
- Cohort 8: Empagliflozin or Dapagliflozin with CVD: A target cohort which includes new users of empagliflozin or dapagliflozin with established CVD for clinical characterization, and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Empagliflozin; Drug: Dapagliflozin
- Cohort 9: DPP-4 inhibitor (i)/ GLP-1 agonist (a)/ other AHA: A comparator cohort which includes new users of any dipeptidyl peptidase-4 (DPP-4) inhibitors, glucagon-like peptide-1 (GLP-1) agonist, or other select antihyperglycemic agents (AHA) for clinical characterization, and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Dipeptidyl Peptidase-4 (DPP-4) Inhibitors; Drug: Glucagon-like Peptide-1 (GLP-1) Agonist; Drug: Anti-hyperglycemic Agents (AHA)
- Cohort 10: DPP-4 (i)/ GLP-1 (a)/ other AHA with CVD: A comparator cohort which includes new users of any DPP-4 inhibitor, GLP-1 agonist, or other select AHA with established CVD for clinical characterization, and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Dipeptidyl Peptidase-4 (DPP-4) Inhibitors; Drug: Glucagon-like Peptide-1 (GLP-1) Agonist; Drug: Anti-hyperglycemic Agents (AHA)
- Cohort 11: DPP-4 (i),GLP-1 (a),TZD, SU, insulin, other AHA: A comparator cohort which includes new users of any DPP-4 inhibitor, GLP-1 agonist, thiazolidinediones (TZD), sulfonylureas (SU), insulin, or other select AHA for clinical characterization, and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Dipeptidyl Peptidase-4 (DPP-4) Inhibitors; Drug: Glucagon-like Peptide-1 (GLP-1) Agonist; Drug: Anti-hyperglycemic Agents (AHA); Drug: Thiazolidinediones (TZD); Drug: Sulfonylureas (SU); Drug: Insulin
- Cohort 12: DPP-4(i), GLP-1(a), TZD, SU, insulin, AHA with CVD: A comparator cohort which includes new users of any DPP-4 inhibitor, GLP-1 agonist, TZD, SU, insulin, or other select AHA with established CVD for clinical characterization, and population-level effect estimation. It will use 4 databases: 1. CCAE 2. MDCR 3. MDCD 4. Optum.
  Interventions: Drug: Dipeptidyl Peptidase-4 (DPP-4) Inhibitors; Drug: Glucagon-like Peptide-1 (GLP-1) Agonist; Drug: Anti-hyperglycemic Agents (AHA); Drug: Thiazolidinediones (TZD); Drug: Sulfonylureas (SU); Drug: Insulin

INTERVENTIONS:
Drug: Canagliflozin — No intervention or treatment assignment imposed by this study. Participants received canagliflozin as a part of routine clinical practice.
  Groups: Cohort 1: Canagliflozin; Cohort 2: Canagliflozin with Cardiovascular Disease (CVD)
Drug: Empagliflozin — No intervention or treatment assignment imposed by this study. Participants received empagliflozin as a part of routine clinical practice.
  Groups: Cohort 3: Empagliflozin; Cohort 4: Empagliflozin with CVD; Cohort 7: Empagliflozin or Dapagliflozin; Cohort 8: Empagliflozin or Dapagliflozin with CVD
Drug: Dapagliflozin — No intervention or treatment assignment imposed by this study. Participants received dapagliflozin as a part of routine clinical practice.
  Groups: Cohort 5: Dapagliflozin; Cohort 6: Dapagliflozin with CVD; Cohort 7: Empagliflozin or Dapagliflozin; Cohort 8: Empagliflozin or Dapagliflozin with CVD
Drug: Dipeptidyl Peptidase-4 (DPP-4) Inhibitors — No intervention or treatment assignment imposed by this study. Participants received DPP-4 inhibitor as a part of routine clinical practice. DPP-4 inhibitors includes: alogliptin, linagliptin, saxagliptin, sitagliptin, vildagliptin.
  Groups: Cohort 10: DPP-4 (i)/ GLP-1 (a)/ other AHA with CVD; Cohort 11: DPP-4 (i),GLP-1 (a),TZD, SU, insulin, other AHA; Cohort 12: DPP-4(i), GLP-1(a), TZD, SU, insulin, AHA with CVD; Cohort 9: DPP-4 inhibitor (i)/ GLP-1 agonist (a)/ other AHA
Drug: Glucagon-like Peptide-1 (GLP-1) Agonist — No intervention or treatment assignment imposed by this study. Participants received GLP-1 agonist as a part of routine clinical practice. GLP-1 agonists includes: albiglutide, dulaglutide, exenatide, liraglutide, lixisenatide.
  Groups: Cohort 10: DPP-4 (i)/ GLP-1 (a)/ other AHA with CVD; Cohort 11: DPP-4 (i),GLP-1 (a),TZD, SU, insulin, other AHA; Cohort 12: DPP-4(i), GLP-1(a), TZD, SU, insulin, AHA with CVD; Cohort 9: DPP-4 inhibitor (i)/ GLP-1 agonist (a)/ other AHA
Drug: Anti-hyperglycemic Agents (AHA) — No intervention or treatment assignment imposed by this study. Participants received other selected AHA as a part of routine clinical practice. Other select AHAs includes: acarbose, bromocriptine, miglitol, nateglinide, repaglinide.
  Groups: Cohort 10: DPP-4 (i)/ GLP-1 (a)/ other AHA with CVD; Cohort 11: DPP-4 (i),GLP-1 (a),TZD, SU, insulin, other AHA; Cohort 12: DPP-4(i), GLP-1(a), TZD, SU, insulin, AHA with CVD; Cohort 9: DPP-4 inhibitor (i)/ GLP-1 agonist (a)/ other AHA
Drug: Thiazolidinediones (TZD) — No intervention or treatment assignment imposed by this study. Participants received TZD as a part of routine clinical practice. TZDs includes: pioglitazone, rosiglitazone, troglitazone.
  Groups: Cohort 11: DPP-4 (i),GLP-1 (a),TZD, SU, insulin, other AHA; Cohort 12: DPP-4(i), GLP-1(a), TZD, SU, insulin, AHA with CVD
Drug: Sulfonylureas (SU) — No intervention or treatment assignment imposed by this study. Participants received SU as a part of routine clinical practice. SUs includes: glipizide, glyburide, glimepiride, chlorpropamide, tolazamide, tolbutamide, acetohexamide
  Groups: Cohort 11: DPP-4 (i),GLP-1 (a),TZD, SU, insulin, other AHA; Cohort 12: DPP-4(i), GLP-1(a), TZD, SU, insulin, AHA with CVD
Drug: Insulin — No intervention or treatment assignment imposed by this study. Participants received Insulin as a part of routine clinical practice.
  Groups: Cohort 11: DPP-4 (i),GLP-1 (a),TZD, SU, insulin, other AHA; Cohort 12: DPP-4(i), GLP-1(a), TZD, SU, insulin, AHA with CVD

SUMMARY:
The primary purpose of study is to estimate the incidence and comparative effect on health outcomes: 1) hospitalization for heart failure, 2) below knee lower extremity amputation. The date of first exposure to the particular drug(s) in the database, where the exposure start is between 1-April-2013 to 15-May-2017 and outcome data for these participants will be analyzed and reported in this study.

ELIGIBILITY:
Inclusion Criteria:

* First exposure to the particular drug(s) in database (index date)
* Exposure start is between 1 April 2013 and 15 May 2017
* At least 365 days of continuous observation time prior to index
* At least 1 condition occurrence of 'Type II diabetes' any time in the prior continuous observation time (which is at least 365 days long) before or on the index date (first exposure to the particular drug(s) in database)

For cohort with 'established cardiovascular disease - At least 1 occurrence of 'conditions indicating established cardiovascular disease' on or any time in the prior continuous observation time (which is at least 365 days long) prior to the index date

Exclusion Criteria:

- Participants with type 1 diabetes or secondary diabetes prior to or on the index date of exposure were excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants diagnosed with type 2 diabetes mellitus (T2DM) and established cardiovascular (CV) disease over a 4-year period 1 April 2013 and 15 May 2017 will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 714582 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Number of Hospitalizations for Heart Failure | Approximately 4-years
  Number of hospital admissions with a primary diagnosis of 'heart failure' will be reported.
Number of Participants with Below Knee Lower Extremity Amputation Events | Approximately 4-years
  Number of participants with new below-knee lower extremity amputation procedures, excluding recent (within 30 day) revisions will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Janssen Investigative Site, Titusville, New Jersey, United States